CLINICAL TRIAL: NCT01662960
Title: Visual Feedback Therapy for Treating Individuals With Hemiparesis Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Steve Jax, Institute Scientist, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HN 4404; NIH R01 HD068565 (Other: Einstein Healthcare Network)
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Hemiparesis; Stroke
Keywords: stroke; hemiparesis; arm movement; sensory functioning
MeSH Terms: conditions — Paresis; Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror therapy (Experimental): 4 weeks of home-based mirror therapy. Participants practiced making movements with mirrored visual feedback of the low-functioning arm.
  Interventions: Behavioral: Mirror therapy
- Divider therapy (Active Comparator): 4 weeks of home-based divider therapy (control therapy to mirror therapy; mirror replaced by a divider). Participants practiced making movements with no visual feedback of the low-functioning arm.
  Interventions: Behavioral: Divider therapy

INTERVENTIONS:
Behavioral: Mirror therapy — A home-based therapy involving mirrored visual feedback
  Arms: Mirror therapy
Behavioral: Divider therapy — A home-based therapy involving removed visual feedback.
  Arms: Divider therapy

SUMMARY:
The purpose of the study is to determine whether an existing treatment for problems that participants have with making movements after a stroke can be performed at home.

DETAILED DESCRIPTION:
This study will compare two forms of home-based treatment for post-stroke problems making movements with the arms and hands. After initial pre-treatment assessments, participants will complete 4 weeks of treatment, with assessments after each week of treatment and 3 months after the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 6 months or more post-stroke
* upper extremity Fugl-Meyer score between 10 and 50
* no longer participating in upper-extremity physical or occupational therapy
* sufficient comprehension ability to understand instructions

Exclusion Criteria:

* previous head trauma, psychiatric illness or chronic exposure to medications that might be expected to have lasting consequences for the central nervous system (e.g., haloperidol, dopaminergics)
* dementia

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jax, Ph. D., Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Einstein Medical Center Elkins Park, Elkins Park, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirror Therapy: High Functioning: 4 weeks of home-based mirror therapy. Participants practiced making movements with mirrored visual feedback of the low-functioning arm.
  High functioning was defined as pre-treatment upper extremity Fugl-Meyer score of 30-50.
- Mirror Therapy: Low Functioning: 4 weeks of home-based mirror therapy. Participants practiced making movements with mirrored visual feedback of the low-functioning arm.
  Low functioning was defined as pre-treatment upper extremity Fugl-Meyer score of 10-29.
- Divider Therapy: High Functioning: 4 weeks of home-based divider therapy (control therapy to mirror therapy; mirror replaced by a divider). Participants practiced making movements with no visual feedback of the low-functioning arm.
  High functioning was defined as pre-treatment upper extremity Fugl-Meyer score of 30-50.
- Divider Therapy: Low Functioning: 4 weeks of home-based divider therapy (control therapy to mirror therapy; mirror replaced by a divider). Participants practiced making movements with no visual feedback of the low-functioning arm.
  Low functioning was defined as pre-treatment upper extremity Fugl-Meyer score of 10-29.
Period: End of 4 Week Treatment Period
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Started | 25 | 23 | 9 | 15
Completed | 24 | 19 | 8 | 15
Not Completed | 1 | 4 | 1 | 0
Period: 3 Month Follow-up
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Started | 24 | 19 | 8 | 15
Completed | 21 | 16 | 5 | 13
Not Completed | 3 | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning | Total
Number analyzed (Participants) | 25 | 23 | 9 | 15 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (12.3) | 53.7 (14.9) | 55.9 (9.7) | 57.5 (12.7) | 57.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 4 | 4 | 25
  Male | 17 | 14 | 5 | 11 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 24 | 22 | 9 | 14 | 69
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 11 | 10 | 4 | 7 | 32
  White | 12 | 12 | 5 | 7 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 3
Upper Extremity Fugl-Meyer [Mean (Standard Deviation); unit: score on a scale] — This test measures impairment-level ability to move the arm and hand. Scores range from 0 to 66, with higher scores indicating greater ability to move the arm and hand.
  score on a scale | 39.1 (6.1) | 17.5 (4.2) | 39.9 (7.8) | 18.8 (6.1) | 28.1 (12.1)
Action Research Arm Test [Mean (Standard Deviation); unit: score on a scale] — The test measures the ability to complete simulated everyday tasks with the arm. Scores range from 0 to 54, with higher scores indicating better performance.
  score on a scale | 36.1 (9.9) | 5.8 (4.4) | 36.3 (13.3) | 6.7 (4.4) | 20.3 (17.1)
Rivermead Assessment of Somatosensory Performance [Mean (Standard Deviation); unit: Proportion of items correct] — This test measures the integrity of sensory perception of the arm. The score is the proportion of items answered correctly, and ranges from 0 to 1 with higher scores indicating better performance.
  Proportion of items correct | 0.72 (0.17) | 0.53 (0.19) | 0.79 (0.20) | 0.56 (0.21) | 0.63 (0.21)
Stroke Impact Scale [Mean (Standard Deviation); unit: score on a scale] — This test measures the self-reported ability to complete everyday tasks with the arm. Total scores for all items are reported. The scale ranged from 0 to 300, with higher scores indicating higher self-reported ability.
  score on a scale | 215.9 (26.4) | 219.9 (35.0) | 226.3 (15.3) | 215.7 (28.7) | 218.4 (30.2)
Wolf Motor Function Test [Mean (Standard Deviation); unit: score on a scale] — The test measures the ability to completed simulated everyday tasks with the arm. The scale ranged from 0 to 75, with higher scores indicating better performance.
  score on a scale | 48.8 (9.5) | 22.7 (5.7) | 50.8 (14.4) | 25.1 (7.2) | 35.8 (15.5)
Virtual-reality Assessment of Navigation [Mean (Standard Deviation); unit: proportion difference] — This test measures the ability to detect lateralized attention problems in a simulated navigation test. Evidence for lateralized attentional problems was defined as a 20% difference in item detection between the left and right side.
  proportion difference | .047 (.051) | .056 (.059) | .022 (.036) | .063 (.086) | .050 (.062)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Fugl-Meyer
Description: This test measures impairment-level ability to move the arm and hand. Scores range from 0 to 66, with higher scores indicating greater ability to move the arm and hand.
Time Frame: Immediately after 1 month of treatment
Population: All participants who started the treatment were included. Data for any participants who failed to complete the treatment were imputed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 25 | 23 | 9 | 15
score on a scale | 43.8 (9.4) | 21.4 (5.7) | 42.8 (8.7) | 21.5 (6.3)
Statistical Analysis 1: Comparison: Mirror Therapy: High Functioning vs Mirror Therapy: Low Functioning vs Divider Therapy: High Functioning vs Divider Therapy: Low Functioning; Test type: Superiority — Test for the superiority of Mirror therapy over Divider therapy; p = .443, ANCOVA — ANCOVA analysis with post-treatment score as the dependent variable, therapy type (Mirror therapy or Divider Therapy) as the independent variable, and pre-treatment score as the covariate. P-value reported is for the main effect of therapy type; Slope = 2.2

2. Primary Outcome: Action Research Arm Test
Description: The test measures the ability to complete simulated everyday tasks with the arm. Scores range from 0 to 54, with higher scores indicating better performance.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 25 | 23 | 9 | 15
score on a scale | 39.9 (11.8) | 7.1 (5.0) | 39.1 (13.6) | 7.7 (5.6)
Statistical Analysis 1: Comparison: Mirror Therapy: High Functioning vs Mirror Therapy: Low Functioning vs Divider Therapy: High Functioning vs Divider Therapy: Low Functioning; Test type: Superiority — Test for the superiority of Mirror therapy over Divider therapy; p = .80, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Slope = 0.4

3. Primary Outcome: Rivermead Assessment of Somatosensory Performance
Description: This test measures the integrity of sensory perception of the arm. The score is the proportion of items answered correctly, and ranges from 0 to 1 with higher scores indicating better performance.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of items correct.
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 25 | 23 | 9 | 15
Proportion of items correct. | 0.76 (0.18) | 0.52 (0.19) | 0.79 (0.18) | 0.60 (0.20)
Statistical Analysis 1: Comparison: Mirror Therapy: High Functioning vs Mirror Therapy: Low Functioning vs Divider Therapy: High Functioning vs Divider Therapy: Low Functioning; Test type: Superiority — Test for the superiority of Mirror therapy over Divider therapy; p = .93, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Slope = -.002

4. Primary Outcome: Virtual-reality Assessment of Navigation
Description: This test measures the ability to detect lateralized attention problems in a simulated navigation test. Evidence for lateralized attentional problems was defined as a 20% difference in item detection between the left and right side.
Time Frame: 1 month
Population: No participants were administered the test in the post-treatment phase because no participant exhibited a baseline 20% difference in item detection between the left and right side.
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Stroke Impact Scale
Description: This test measures the self-reported ability to complete everyday tasks with the arm. Total scores for all items are reported. The scale ranged from 0 to 300, with higher scores indicating higher self-reported ability.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 25 | 23 | 9 | 15
score on a scale | 221.0 (32.5) | 231.6 (43.7) | 237.8 (25.7) | 217.0 (26.7)
Statistical Analysis 1: Comparison: Mirror Therapy: High Functioning vs Mirror Therapy: Low Functioning vs Divider Therapy: High Functioning vs Divider Therapy: Low Functioning; Test type: Superiority — Test for the superiority of Mirror therapy over Divider therapy; p = .28, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Slope = 10.7

6. Secondary Outcome: Wolf Motor Function Test
Description: The test measures the ability to completed simulated everyday tasks with the arm. The scale ranged from 0 to 75, with higher scores indicating better performance.
Time Frame: 1 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
Number analyzed (Participants) | 25 | 23 | 9 | 15
score on a scale | 50.0 (10.0) | 22.3 (6.0) | 50.4 (13.8) | 24.7 (6.7)
Statistical Analysis 1: Comparison: Mirror Therapy: High Functioning vs Mirror Therapy: Low Functioning vs Divider Therapy: High Functioning vs Divider Therapy: Low Functioning; Test type: Superiority — Test for the superiority of Mirror therapy over Divider therapy; p = .86, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Slope = -.36

ADVERSE EVENTS:
Time Frame: From Baseline screening until 3-month post-treatment follow-up.
Arm/Group | Mirror Therapy: High Functioning | Mirror Therapy: Low Functioning | Divider Therapy: High Functioning | Divider Therapy: Low Functioning
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/9 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/9 | 0/15
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 0/9 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT01662960/Prot_SAP_000.pdf